CLINICAL TRIAL: NCT02162264
Title: Post-marketing Surveillance of Donepezil Hydrochloride -Investigation of the Factors That Affect Aricept Medication Persistence Rate and the Safety and Efficacy in Patients With Alzheimer's Disease in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: ART08T
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; donepezil hydrochloride
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- E2020
  Interventions: Drug: Donepezil Hydrochloride

INTERVENTIONS:
Drug: Donepezil Hydrochloride — Initial dose of 3 mg orally once daily. After 1-2 weeks, dosage increased to 5 mg orally once daily. After 4 or more weeks, dosage increased to 10 mg orally once daily for patients with severe dementia of Alzheimer's type. Dose reduced appropriately according to patient's symptoms.
  Other Names: Aricept

SUMMARY:
To investigate the factors that affect Aricept medication persistence rate and the safety and efficacy in patients with Alzheimer's Disease in clinical practice

ELIGIBILITY:
Inclusion criteria:

Patients diagnosed with Alzheimer's Disease and administered Aricept for the first time.

Exclusion criteria:

Patients with a history of hypersensitivity to any ingredients of Aricept or piperidine derivatives.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Alzheimer's Disease
Sampling Method: Non-Probability Sample
Enrollment: 8662 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2016-07-22 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in the Mini-Mental State Examination (MMSE) Score | Baseline, Month 3, Month 6, and Month 12

SECONDARY OUTCOMES:
Investigations on adverse events and adverse drug reactions | Baseline and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Omata, Study Director — Drug Fostering and Evolution Coordination Department, Eisai Co., Ltd.
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Result] Geriatric Medicine 55(10): 1131-1145, 2017.